CLINICAL TRIAL: NCT04499235
Title: Double-Blind, Randomized, Placebo-Controlled Trial of AKST4290 for Adjunctive Treatment of Mild to Moderate Bullous Pemphigoid
Brief Title: A Study to Assess the Therapeutic Effect and Safety of Adjunctive AKST4290 in Subjects With Bullous Pemphigoid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated by the Sponsor due to operational challenges stemming from the coronavirus disease 2019 (COVID-19) pandemic, treatment limitations, rarity of the disease, and drug supply considerations.
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AKST4290-221
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Pemphigoid, Bullous
Keywords: Autoimmune disease; Skin disease; Vesiculobullous
MeSH Terms: conditions — Pemphigoid, Bullous; Autoimmune Diseases; Skin Diseases | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mometasone furoate + AKST4290 (Experimental): Subjects will receive mometasone furoate concurrently with AKST4290, 400 mg twice daily, until disease control is reached.
  Interventions: Drug: Mometasone furoate; Drug: AKST4290
- Mometasone furoate + Placebo (Placebo Comparator): Subjects will receive mometasone furoate concurrently with placebo until disease control is reached.
  Interventions: Drug: Mometasone furoate; Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate — Topical mometasone furoate
Drug: AKST4290 — Oral AKST4290
  Arms: Mometasone furoate + AKST4290
Drug: Placebo — Oral placebo
  Arms: Mometasone furoate + Placebo

SUMMARY:
This study will evaluate the therapeutic effect and safety of adjunctive AKST4290 in subjects with bullous pemphigoid (BP).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the therapeutic effect and safety of adjunctive AKST4290 in subjects with bullous pemphigoid (BP). Subjects will receive topical mometasone furoate cream (MFC) therapy concurrently with study agent (placebo or AKST4290) in an inpatient setting until disease control is reached (duration of inpatient stay is dependent upon individual disease course, but is estimated between 1-3 weeks).

Subjects will receive rescue therapy at any time if their clinical condition worsens or if their clinical condition fails to improve by the completion of Week 1 on study treatment, as assessed by the investigator. Rescue therapy will consist of whole-body clobetasol propionate cream (CPC) (15-50g) and/or oral prednisone (0.5 mg/kg per day), as determined by the investigator. Subjects who receive rescue therapy will remain in the study until disease control, unless they are withdrawn or withdraw from participation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate BP at screening.
* Treatment naïve or initiation of whole-body high potency topical steroid treatment ≤ 7 days of screening (lesion-only treatment for any amount of time with any topical steroids prior to screening is allowed without restriction).
* Provide a signed and dated informed consent form in accordance with local regulations and/or IRB/IEC guidelines.

Exclusion Criteria:

* Severe BP.
* Initiation of gliptins and other treatments (e.g., etanercept, sulfasalazine, furosemide, penicillin) that can trigger BP if this treatment was started within 4 weeks prior to screening and is considered possibly related to the onset of BP.
* Any concomitant medications in the last 3 months prior to screening and assessed by the investigator as possibly related to the development of BP.
* Planned use of intravenous immunoglobulin or other concomitant treatments for BP (i.e., doxycycline, dapsone) during the study period.
* Use of systemic immunosuppressants (i.e., mycophenolate, azathioprine, methotrexate) within 4 weeks prior to screening.
* Treatment with rituximab within 1 year prior to screening.
* Subjects taking warfarin.
* Use of systemic steroids (>10 mg prednisone or equivalent/day) within 14 days of first dose of study agent or known diseases (other than BP) that could require the use of systemic steroids within the study period.
* Clinically relevant abnormal laboratory value at screening, including hematology, blood chemistry, or urinalysis (laboratory testing may be repeated once during the screening phase).
* Participation in studies of investigational drugs must have been discontinued within 30 days or 5 half lives of the drug (whichever was longer) prior to screening.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (8):
- Germany (8):
  - Universitätsklinikum Carl Gustav Carus Dresden Klinik und Poliklinik für Dermatologie, Dresden
  - Universitätsklinikum Düsseldorf Klinik für Dermatologie, Düsseldorf
  - Universitätsklinikum Erlangen - Hautklinik, Erlangen
  - Universitätsklinikum Freiburg Klinik für Dermatologie und Venerologie, Freiburg im Breisgau
  - Universitätsklinikum Schleswig-Holstein Klinik für Dermatologie, Allergologie und Venerologie (Hautklinik) Exzellenzzentrum Entzündungsmedizin, Lübeck
  - Universitätsklinikum Magdeburg A.ö.R. Universitätshautklinik, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz Hautklinik Clinical Research Center (CRC), Mainz
  - Universitätsklinikum Würzburg Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Würzburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants per the protocol are participants who are randomized to mometasone furoate + AKST4290 or mometasone furoate + placebo. Subjects screened but not randomized are not reflected in Participant Flow. The study enrolled 6 subjects of the planned 30 subjects before study prematurely terminated by the Sponsor.
Period: Overall Study
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7.78) | 60 | 65 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Achieve Disease Control Without Rescue Therapy
Description: Disease control is defined as ≤ 3 new blisters/eczematous lesions/urticarial plaques/day and healing of existing blisters/eczematous lesions/urticarial plaques without requiring rescue therapy.
Time Frame: Baseline to up to 3 weeks (until disease control)
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 5 | 1
Participants | 2 | 1

2. Secondary Outcome: Number of Participants With TEAEs, Assessed by Seriousness and Severity
Description: Treatment-emergent AEs summarized by MedDRA coding terms; separate tabulations produced for incidence, seriousness and severity of AEs
Time Frame: Baseline to 5 weeks
Population: The Safety Evaluable Set includes all randomized subjects who receive at least 1 dose of the study agent (AKST4290 or placebo)
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 5 | 1
Participants
  Subjects Reporting at Least One TEAE | 2 | 1
  Subjects Reporting at Least One Serious TEAE | 0 | 1
  TEAE by Severity: Mild | 2 | 0
  TEAE by Severity: Moderate | 0 | 0
  TEAE by Severity: Severe | 0 | 1

3. Secondary Outcome: Time to Disease Control
Description: Time to disease control by treatment day/week. The time to disease control is calculated as the date of disease control minus Date of Visit 2 (Baseline (Day 1)) plus 1.
Time Frame: Baseline to up to 3 weeks (until disease control)
Population: Analysis population includes subjects who achieved disease control with and without rescue therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 5 | 1
Participants
  Time (Days) to Disease Control: 8 | 1 | 0
  Time (Days) to Disease Control: 11 | 2 | 0
  Time (Days) to Disease Control: 15 | 0 | 1
  Time (Days) to Disease Control: 16 | 1 | 0
  Time (Days) to Disease Control: 22 | 1 | 0

4. Secondary Outcome: Time to Rescue Therapy
Description: Time to rescue therapy by treatment day/week. The time to rescue therapy is calculated as the start date of the first rescue therapy minus Date of Visit 2 (Baseline (Day 1)) plus 1.
Time Frame: Baseline to up to 3 weeks (EOT). EOT occurs at disease control (assessed every day from Week 1/Day 7 up to Week 3/Day 21 +/- 2 days) or at Week 3/Day 21 +/- 2 days when the subject is discontinued from treatment due to not reaching disease control.
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 5 | 1
Participants
  Time (Days) to Rescue Therapy: 4 | 1 | 0
  Time (Days) to Rescue Therapy 8 | 1 | 0
  Time (Days) to Rescue Therapy 9 | 1 | 0

5. Secondary Outcome: The Bullous Pemphigoid Disease Area Index (BPDAI) Score
Description: Change from baseline in BPDAI score at End of Treatment (EOT). Subscales for the BPDAI include the skin blister score (range 0-120), skin urticarial score (range 0-120), mucosal activity score (range 0-120), and damage score (range 0-12). Higher scores indicate greater disease activity or damage.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 5 | 1
score on a scale
  Total BPDAI Skin Blister Score: Baseline | 15 (12.83) | 13.0
  Total BPDAI Skin Blister Score: EOT | 7.4 (7.02) | 8.0
  Total BPDAI Skin Urticarial Score: Baseline | 16.4 (9.15) | 14.0
  Total BPDAI Skin Urticarial Score: EOT | 9.2 (6.38) | 12.0
  Total BPDAI Mucosal Activity Score: Baseline | 3.4 (7.60) | 0
  Total BPDAI Mucosal Activity Score: EOT | 1.6 (3.58) | 0
  Total BPDAI Damage Score: Baseline | 5.0 (4.18) | 9.0
  Total BPDAI Damage Score: EOT | 5.0 (3.81) | 8.0

6. Secondary Outcome: The Bullous Pemphigoid Disease Area Index Visual Analog Scale (BPDAI-VAS)
Description: Change from baseline in pruritus as evaluated by the BPDAI-VAS at End of Treatment (EOT). EOT occurs at disease control (up to 3 weeks) or at Week 3 when the subject is discontinued from treatment due to not reaching disease control. Scores for the BPDAI-VAS can range from 0 to 30, with higher scores indicating a worse condition.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 5 | 1
score on a scale
  BPDAI-VAS Baseline | 19.4 (5.68) | 15.0
  BPDAI-VAS EOT | 9.2 (3.42) | 4.0

7. Secondary Outcome: Total Cumulative Steroid Exposure
Description: Total cumulative steroid exposure (cortisol equivalent/kg) by treatment group
Time Frame: as for outcome 4
Population: Total cumulative steroid exposure is calculated based on oral route treatment from Day 1 to EOT/disease control. Subjects with no oral route treatment were excluded from analysis.
Measure: Mean (Standard Deviation); unit: mg cortisol equivalent/kg
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 3 | 0
mg cortisol equivalent/kg | 260 (210) |

8. Secondary Outcome: Maximum Daily Steroid Dose
Description: Evaluation of maximum daily steroid dose at baseline, by treatment week, and at disease control. Study Day 1 is defined as the initiation of study treatment. 1 mg/kg prednisolon(e) = 5 mg/kg cortisone.
Time Frame: as for outcome 4
Population: The analysis population includes subjects who received systemic steroids. In the AKST4290 group, 3 subjects received systemic steroids. In the Placebo group, the single subject did not have systemic steroid exposure.
Measure: Number; unit: mg cortisol equivalent/kg
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
Number analyzed (Participants) | 3 | 0
mg cortisol equivalent/kg
  Maximum Daily Steroid Dose Occurred: Day 4: number analyzed (Participants) | 1 | 0
  Maximum Daily Steroid Dose Occurred: Day 4 | 175 |
  Maximum Daily Steroid Dose Occurred: Day 8: number analyzed (Participants) | 1 | 0
  Maximum Daily Steroid Dose Occurred: Day 8 | 150 |
  Maximum Daily Steroid Dose Occurred: Day 11: number analyzed (Participants) | 1 | 0
  Maximum Daily Steroid Dose Occurred: Day 11 | 150 |

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Mometasone Furoate + AKST4290 | Mometasone Furoate + Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/1
Other Adverse Events (participants affected / at risk) | 2/5 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate + AKST4290 (N=5) | Mometasone Furoate + Placebo (N=1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate + AKST4290 (N=5) | Mometasone Furoate + Placebo (N=1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement contains language that restricts the PI from discussing or publishing Sponsor confidential and/or proprietary information. The embargo period may be extended by mutual agreement of the Sponsor and PI.

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT04499235/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT04499235/SAP_001.pdf